CLINICAL TRIAL: NCT01662206
Title: Probiotics (Lactobacillus Gasseri, Bifidobacterium Bifidum, Bifidobacterium Longum) on Immune and Intestinal Health in Healthy Older Adults
Brief Title: Probiotics (L. Gasseri, B. Bifidum, B. Longum) on Immune and Intestinal Health in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 236-2012; 236-2012 (Other Grant/Funding Number: Wakunaga of America Co., Ltd.)
Record Dates: First submitted 2012-07-26; First posted 2012-08-10 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: adults; probiotics; immune function; microbiota; digestive health
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Capsules containing Lactobacillus gasseri, Bifidobacterium bifidum, and Bifidobacterium longum
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Capsules containing placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 2 capsules daily containing Lactobacillus gasseri, Bifidobacterium bifidum and Bifidobacterium longum (1.5 billion cells per capsule prior to expiration)
  Arms: Probiotic
Dietary Supplement: Placebo — 2 capsules daily containing 348.25 mg of potato starch
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether healthy older adults, aged 65 to 80 years, consuming a probiotic each day for three weeks will have improved immune strength and digestive health. It is hypothesized that older adults consuming the probiotics will see a shift in their microbiota towards the "healthy" bacteria resulting in a greater proportion of immune cells, decreased inflammation, and better digestive health.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled crossover design with two 3-week interventions and a 5-week washout period in between. Thirty-six participants will be enrolled. With informed consent, the daily questionnaire will be administered and a baseline stool sample will be obtained during the week before the start of each intervention period. Blood and saliva will be collected on the first and last day of each intervention period to assess immune function. A final stool sample will be obtained in the last week of the intervention period. Nutritional status, which can impact immune function, will be assessed using the Mini-Nutritional Assessment, Block Fiber Screen, and the Block 2005 Food Frequency Questionnaire. Daily questionnaires will record intake of the probiotic or placebo, level of stress, hours of sleep, visits to the physician, new medications, number of stools, etc. The Gastrointestinal Symptom Response Scale, which records gastrointestinal symptoms, such as bloating, gas, diarrhea, and constipation, over the past week will be completed at baseline and weekly during the interventions and the week following the interventions.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 80 years of age.
* willing and able to complete the Informed Consent Form in English
* willing to provide demographic information (age, race)
* willing and able to complete daily and weekly questionnaires regarding general wellness, bowel function and gastrointestinal symptoms.
* willing to provide 4 blood, 4 stool, and 4 saliva samples
* willing to discontinue any immune-enhancing dietary supplements ( e.g., prebiotics supplements, Echinacea, fish oil, vitamin E >200% of the RDA).
* able to take the study probiotic without the aid of another person.

Exclusion Criteria:

* not meet the above criteria.
* taking any medication for constipation or diarrhea.
* currently taking any anti-inflammatory drugs on a regular basis.
* current smoker.
* typically consume fermented foods or probiotics (e.g., yogurts with live, active cultures or supplements).
* currently being treated for or have any of the following physician- diagnosed diseases or conditions: HIV/AIDS, immune modulating diseases (autoimmune, hepatitis, cancer, etc.), kidney disease, diabetes or gastrointestinal disease or conditions (such as ulcerative colitis, Crohn's disease, gastroparesis, cancer, peptic ulcer disease, Celiac disease, short bowel disease, ileostomy, colostomy) other than GERD or diverticular disease or have a central venous catheter.
* received chemotherapy or other immune suppressing therapy within the last year.
* received antibiotic therapy in the past two months.
* cannot schedule planned immunizations to at least 4 weeks before the start of the study, in the week following the second blood draw, or after the 4th blood draw.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in cytokine production | Measured at baseline and after 3 weeks of supplementation for each arm
  Peripheral blood mononuclear cell cytokine production following lipopolysaccharide stimulation
Change in bacterial species measured in fecal samples | Measured at baseline and after 3 weeks of supplementation for each arm
  * Microbial diversity measured by 454 16S rRNA sequence analysis
  * qPCR to quantify changes in bacteria of interest

SECONDARY OUTCOMES:
Change in digestive symptoms on the Gastrointestinal Symptom Response Scale | Measured at baseline, weeks 1, 2, 3 and 4 of each arm
  Symptoms (gas, bloating, diarrhea, etc.) reported on a daily questionnaire and a weekly Gastrointestinal Symptom Response Scale
Change in Mucosal immune function | Measured at baseline and after 3 weeks of supplementation for each arm
  sIgA

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States